CLINICAL TRIAL: NCT05112367
Title: Retrospective Study on the Management of Pediatric Anaphylaxis and Clinical Signs of Allergy in the Pediatric Emergency Department of Montpellier University Hospital
Brief Title: Epidemiology and Management of Pediatric Anaphylaxis and Allergy in the Pediatric Emergency Department of Montpellier
Acronym: Ana-Ped
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0613
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Anaphylaxis; Allergy
Keywords: Children; Emergency; Epinephrine
MeSH Terms: conditions — Anaphylaxis; Hypersensitivity; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anaphylaxis is a severe life-threatening reaction following exposure to an antigen. Its incidence is progressively increasing in the general population over years, especially among children. The diagnosis can be difficult, and recommendations for follow up and prescription for an emergency kit are rarely provided after emergency visit. The Investigators will evaluate the management of pediatric anaphylaxis and clinical signs of allergy in the pediatric emergency department of Montpellier University Hospital

ELIGIBILITY:
Inclusion criteria:

* Patients evaluated at the Montpellier University Hospital, Allergy Unit ;
* Children consulting for suspected allergy from 2016 to 2020

Exclusion criteria:

- Patients under legal protection, under guardianship or under curatorship;

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children consulting in the paediatric emergency department of Montpellier for suspected allergy from 2016 to 2020
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the management of pediatric anaphylaxis of allergy | day 1
  Evaluation of the management of pediatric anaphylaxis of allergy in the pediatric emergency department of Montpellier University Hospital.
Evaluation of the management of pediatric clinical signs evocative of allergy in the pediatric emergency department of Montpellier University Hospital. | day 1
  Evaluation of the management of pediatric clinical signs evocative of allergy in the pediatric emergency department of Montpellier University Hospital.

SECONDARY OUTCOMES:
Evaluation of an appropriate use of epinephrine | day 1
  Evaluation of an appropriate use of epinephrine
Evaluation of an appropriate use of a possible follow-up of patients after the episode | day 1
  Evaluation of an appropriate use of a possible follow-up of patients after the episode

CONTACTS AND LOCATIONS:
Overall Officials: Davide CAIMMI, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Clark E, Kase Tanno L, Vo T, Blanc B, Demoly P, Caimmi D. Anaphylaxis management in a French pediatric emergency department: Lessons from the ANA-PED study. Clin Transl Allergy. 2023 Aug;13(8):e12289. doi: 10.1002/clt2.12289. PMID 37632240